CLINICAL TRIAL: NCT03493776
Title: Safety and Immunogenicity of Non-live, Recombinant Subunit Herpes Zoster Vaccine Before and After Lung Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deepali Kumar (Other)
Responsible Party: Sponsor-Investigator, Deepali Kumar, MD, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHN-Shingrix-001
Record Dates: First submitted 2018-03-29; First posted 2018-04-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Varicella Zoster Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-Transplant Group (Active Comparator): VZV Subunit vaccine will be administered
  Interventions: Biological: VZV subunit vaccine
- Post-Transplant Group (Experimental): VZV Subunit vaccine will be administered
  Interventions: Biological: VZV subunit vaccine

INTERVENTIONS:
Biological: VZV subunit vaccine — VZV subunit vaccine

SUMMARY:
The investigators plan to study the immunogenicity of the vaccine before and after lung transplantation. Patients (at least 50 years old) before and after lung transplantation will be enrolled. The investigators hypothesize that the recombinant varicella-zoster subunit vaccine is able to induce cellular immunogenicity after transplantation.

DETAILED DESCRIPTION:
Solid organ transplant recipients receive lifelong immunosuppression and are at increased risk for reactivation of all herpesviruses including VZV. Epidemiologic studies show the cumulative incidence in lung transplant recipients of reactivation to be 15-20%. A non-live, recombinant subunit vaccine (Shingrix; GSK vaccines) was recently licensed for the prevention of shingles in people aged 50 years or older. The investigators plan to study the immunogenicity of the vaccine before and after lung transplantation. Patients (at least 50 years old) before and after lung transplantation will be enrolled. The investigators hypothesize that the recombinant varicella-zoster subunit vaccine is able to induce cellular immunogenicity after transplantation.

ELIGIBILITY:
Inclusion Criteria Post-Transplant Vaccine Group:

* Single or double lung transplant recipient.
* Age ≥50 years

Exclusion Criteria Post-Transplant Vaccine Group:

* Has already received varicella zoster subunit vaccine in the past
* Shingles within the last 12 months
* Ongoing CMV viremia > 200 IU/mL
* HIV infection
* Diagnosis of malignancy (eg PTLD)

Inclusion Criteria Pre-Transplant Vaccine Group:

* On waiting list for lung transplantation
* Age ≥50 years

Exclusion Criteria Pre-Transplant Vaccine Group:

* Has already received Shingrix or Zostavax (live shingles vaccine) in the past
* Systemic prednisone ≥20 mg per day (or equivalent dose of any corticosteroid)
* Other (than prednisone < 20mg per day or equivalent dose of any corticosteroid) systemic immunosuppressive therapy such as mycophenolate or tacrolimus
* Shingles within the last 12 months
* HIV infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Cellular immunity to varicella zoster induced by varicella zoster subunit vaccine. | 4 weeks after second dose of vaccine
  Cellular immunogenicity against VZV induced by varicella zoster subunit vaccine in lung transplant recipients measured as a percentage of CD4+ and CD8+ T-cells measured by intracellular flow-cytometry based staining. The cellular immunogenicity of the vaccine in lung transplant recipients will be compared to the control group (pre-transplant vaccination).

SECONDARY OUTCOMES:
Humoral immunogenicity to varicella zoster induced by varicella zoster subunit vaccine in lung transplant recipients. | 4 weeks after second dose of vaccine
  Humoral immunogenicity (increase of GMTs of anti-VZV antibodies) in lung transplant
Humoral immunogenicity to varicella zoster induced by varicella zoster subunit vaccine in post-transplant group vs. pre-transplant group | 4 weeks after second dose of vaccine
  Humoral immunogenicity (GMTs of anti-VZV antibodies compared pre and post vaccination) against VZV induced by varicella zoster subunit vaccine in lung transplant recipients compared to the pre-transplant control group.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — Multi organ transplant program, University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No